CLINICAL TRIAL: NCT02573909
Title: The Safety and Efficacy of Epidural Oxycodone
Acronym: epioksipanu
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Admescope Ltd (Industry)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH2014-004313-82
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: similar syringes equal amount of drug
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone intravenously (Experimental): Oxycodone 0,1 mg/kg IV
  Interventions: Drug: Oxycodone epidurally
- Oxycodone epidurally (Experimental): Oxycodone 0,1 mg/kg epidurally
  Interventions: Drug: Oxycodone intravenously

INTERVENTIONS:
Drug: Oxycodone intravenously — Oxycodone intravenously 0,1mg/kg
  Other Names: oxycodoneIV
  Arms: Oxycodone epidurally
Drug: Oxycodone epidurally — Oxycodone 0,1 mg epidurally
  Other Names: oxycodoneEpid
  Arms: Oxycodone intravenously

SUMMARY:
There are conflicting results in earlier studies concerning the safety and efficacy of epidural oxycodone. In a study by Bäcklund and colleagues, epidural oxycodone was as effective as intravenous oxycodone, so they did not recommend epidural use of oxycodone. In another study, Yanagidate and Dohi reported that oxycodone was as effective in pain treatment with double dose compared to epidural morphine. In our previous study, epidural oxycodone provided safe and effective pain relief when compared to intravenous oxycodone.

In the present study, the aim was to compare the efficacy and safety of epidural or intravenous oxycodone in patients undergoing elective gynecological surgery with planned epidural pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* Planned gynecological lower abdomen surgery with epidural pain treatment
* Informed consent obtained

Exclusion Criteria:

* Planned surgery under regional anesthesia
* contraindication to the study drug
* contraindication to the lumbar puncture
* Contraindication to oxycodone
* Pregnancy or lactation
* no informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
amount of rescue medicine | from zero hours up to four hours
  The amount of rescue pain medication given after study drug administration up to four hours

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, PhD, Principal Investigator — Kuopio University Hospital, Kuopio, Finland
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Undecided